CLINICAL TRIAL: NCT02648802
Title: Cavity Shaving in Breast Conserving Surgery With Intraoperative Cavity Margin Assessment: A Single Center,Randomized,Controlled Trial
Brief Title: Cavity Shaving in Breast Conserving Surgery for Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Fengxi Su, Director of the Breast Tumor Department of Sun Yat-Sen Memorial Hospital, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSBCS1
Record Dates: First submitted 2016-01-03; First posted 2016-01-07 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
Keywords: breast-conserving surgery(BCS); Cavity shave margin; Proportion of positive margins
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cavity shaving and CM assessment (Experimental): Standardized BCS with additional cavity shaving before CM assessment.
  Interventions: Procedure: Cavity shaving; Procedure: Standardized BCS+CM assessment.
- CM assessment (Placebo Comparator): Standardized BCS with CM assessment.
  Interventions: Procedure: Standardized BCS+CM assessment.

INTERVENTIONS:
Procedure: Cavity shaving — Resect the residual cavity circumferentially (superior, inferior, medial, lateral) and the thickness of the cavity shaving depends on the surgeon's discretion (Recommended 0.5-1.0cm). The principles of the cavity shaving includes: 1) do not compromise the cosmetic outcomes; 2) covers the entire cavity;
  Arms: Cavity shaving and CM assessment
Procedure: Standardized BCS+CM assessment. — For standardized BCS(Chen K, et al. Ann Surg Oncol. 2012), we resect a rim of 1 cm macroscopically normal tissue around the tumor. The anterior and posterior margins of the tumor-containing specimen extended up to the subdermal plane of the skin and down to the pectoralis major fascia, respectively. The anterior and posterior CMs assessment will not be needed. A surgical blade was used for resecting the CMs (superior, inferior, medial and lateral) to render the thickness of the CMs as thin as possible. No procedures were required for distinguishing the inner and outer surface. They were then frozen and cut parallel, but not perpendicular to the largest surface area. CMs were defined as positive when in situ or invasive carcinoma was found intraoperatively by frozen-section analysis.

SUMMARY:
This randomized controlled trial is to evaluate the impact of additional cavity shaving (CS) on pathological cavity margin (CM) status in breast cancer patients. Patients receiving standard breast-conserving surgery (BCS) will be randomized to intra-operative CM assessment versus intra-operative CS followed by CM assessment. The primary objective of this study is to assess the impact of CS on intra-operative CM status, intra-operative re-excision rate, post-operative CM status and re-excision rate, cosmetic outcomes, and on intraoperative time and medical costs.

DETAILED DESCRIPTION:
After stratified and blocked randomization, the patients' name, admission ID and treatment assignment will be written on a slip of paper, and will be placed in a sealed envelop. A label with the patients' name and admission ID will be placed on the sealed envelop, which will be kept in a locked file. On the day of surgery, a research coordinator will bring the sealed envelope to the operation room. During the standard-of-care BCS, the tumor was excised with a rim of grossly normal tissue. Additional resections are allowed when any of the margins of the tumor-containing specimen were suspected to be inadequate on the basis of standard gross evaluation by surgeons. Prior to intra-operative CM assessment, the research co-ordinator will unseal the envelop and determine which procedure has been designated to the patient. The cosmetic outcome and the quality of life will be evaluated at the day of discharge, after completion of radiotherapy and one year by the patient herself, her partner and a research co-ordinator.

ELIGIBILITY:
Inclusion Criteria:

* Female
* At least 18 years of age and no more than 65 years of age
* Able to understand and willing to sign an informed consent document
* Willing and planning to undergo the breast-conserving surgery
* ECOG≤ 2

Exclusion Criteria:

* Inflammatory breast cancer
* Preference for mastectomy instead of breast-conserving surgery
* Necessity to undergo oncoplastic breast surgery
* Prior surgical treatment, including ultrasound-guided vacuum-assisted biopsy and excision biopsy.
* Prior systemic therapy for this diagnosis, including neoadjuvant chemotherapy, neoadjuvant endocrine therapy.
* History of prior breast/axillary radiation therapy
* Known metastatic disease
* Diagnosed as bilateral breast cancer or DCIS
* History of other malignancy ≤ 5 years previous
* Preoperation evaluation indicates tumor size>5cm
* Preoperation evaluation indicates multicenter or multifocal breast cancer(including suspicious calcification on mammography)
* Undergoing other clinical trials
* With sever liver disfunction(Child-Pugh C)
* With sever cardiac insufficiency
* With sever renal disfunction
* Pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Positivity rate of CMs by intraoperative frozen section analysis. | Completion of surgery for all enrolled patients (approximately 12 months)
  Proportion of patients with at least one positive(invasive carcinoma or carcinoma in situ, excluding LCIS) CMs on intraoperative frozen section analysis

SECONDARY OUTCOMES:
Intra-operative rate of suspected/positive CM | Completion of surgery for all enrolled patients (approximately 12 months)
  Proportion of patients with at least one positive(invasive carcinoma or carcinoma in situ, excluding LCIS) or suspected CMs on intraoperative frozen section analysis. Suspected CMs were defined as CMs with severe atypical hyperplasia observed by frozen section analysis.
Rate of intra-operative re-excision for suspected/positive CMs | Completion of surgery for all enrolled patients (approximately 12 months)
  For patients with positive CMs, intra-operative re-excision was required. For patients with suspected CMs,intra-operative re-excision is left to the surgeon's discretion
Rate of a second-time surgery for post-operative positive CMs | Completion of surgery for all enrolled patients (approximately 12 months)
  Positive CMs by post-operative pathological analysis may require a second-time surgery for re-excision.
Proportion of patients successfully undergone BCT | Completion of surgery for all enrolled patients (approximately 12 months)
Cost-effectiveness of cavity shaving in BCS as measured by operative time of the surgery | Completion of surgery for all enrolled patients (approximately 12 months)
  Surgery time(start from making the incision to closure) will be analyzed.
Cost-effectiveness of cavity shaving in BCS as measured by medical cost of the surgery | Completion of surgery for all enrolled patients (approximately 12 months)
  Medical costs will be analyzed.
Cosmetic outcome | One year after surgery.
  Patients', partners' and physicians' perceptions of the cosmetic outcomes as measured by Harvard/NSABP/RTOG criteria
Adverse events | One year after surgery.
Quality of life. | One year after surgery.
  Chinese version of validated QLQ-C30 and QLQ-BR23 questionnaire

OTHER OUTCOMES:
Volume of cavity shaving tissue. | Completion of surgery for all enrolled patients (approximately 12 months)
  Water displacement method was used to measure the volume of the tissue resected by cavity shaving.
Weight of cavity shaving tissue. | Completion of surgery for all enrolled patients (approximately 12 months)
Relationship between the volume of tissue excised in association aesthetic outcomes | Completion of surgery for all enrolled patients (approximately 12 months)
  Volume of the excised tissue, including the tumor-containing specimen will be analyzed.
Risk factors for positive CMs | Completion of surgery for all enrolled patients (approximately 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Fengxi Su, M.D., Principal Investigator — Breast Tumor Center, Sun Yat-sen Memorial Hospital, Sun Yat-sen University.
Locations (1):
- Sun-Yat-Sen Memorial Hospital of Sun-Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data will be available after the research paper has been published.

REFERENCES:
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Background] Veronesi U, Cascinelli N, Mariani L, Greco M, Saccozzi R, Luini A, Aguilar M, Marubini E. Twenty-year follow-up of a randomized study comparing breast-conserving surgery with radical mastectomy for early breast cancer. N Engl J Med. 2002 Oct 17;347(16):1227-32. doi: 10.1056/NEJMoa020989. PMID 12393819
- [Background] Moran MS, Schnitt SJ, Giuliano AE, Harris JR, Khan SA, Horton J, Klimberg S, Chavez-MacGregor M, Freedman G, Houssami N, Johnson PL, Morrow M. Society of Surgical Oncology-American Society for Radiation Oncology consensus guideline on margins for breast-conserving surgery with whole-breast irradiation in stages I and II invasive breast cancer. Int J Radiat Oncol Biol Phys. 2014 Mar 1;88(3):553-64. doi: 10.1016/j.ijrobp.2013.11.012. PMID 24521674
- [Background] Morrow M, Jagsi R, Alderman AK, Griggs JJ, Hawley ST, Hamilton AS, Graff JJ, Katz SJ. Surgeon recommendations and receipt of mastectomy for treatment of breast cancer. JAMA. 2009 Oct 14;302(14):1551-6. doi: 10.1001/jama.2009.1450. PMID 19826024
- [Background] Cendan JC, Coco D, Copeland EM 3rd. Accuracy of intraoperative frozen-section analysis of breast cancer lumpectomy-bed margins. J Am Coll Surg. 2005 Aug;201(2):194-8. doi: 10.1016/j.jamcollsurg.2005.03.014. PMID 16038815
- [Background] Chagpar AB, Killelea BK, Tsangaris TN, Butler M, Stavris K, Li F, Yao X, Bossuyt V, Harigopal M, Lannin DR, Pusztai L, Horowitz NR. A Randomized, Controlled Trial of Cavity Shave Margins in Breast Cancer. N Engl J Med. 2015 Aug 6;373(6):503-10. doi: 10.1056/NEJMoa1504473. Epub 2015 May 30. PMID 26028131
- [Background] Kayar R, Civelek S, Cobanoglu M, Gungor O, Catal H, Emiroglu M. Five methods of breast volume measurement: a comparative study of measurements of specimen volume in 30 mastectomy cases. Breast Cancer (Auckl). 2011 Mar 27;5:43-52. doi: 10.4137/BCBCR.S6128. PMID 21494401
- [Background] Chen K, Zeng Y, Jia H, Jia W, Yang H, Rao N, Song E, Cox CE, Su F. Clinical outcomes of breast-conserving surgery in patients using a modified method for cavity margin assessment. Ann Surg Oncol. 2012 Oct;19(11):3386-94. doi: 10.1245/s10434-012-2331-5. Epub 2012 Apr 10. PMID 22488098
- [Derived] Chen K, Zhu L, Chen L, Li Q, Li S, Qiu N, Yang Y, Su F, Song E. Circumferential Shaving of the Cavity in Breast-Conserving Surgery: A Randomized Controlled Trial. Ann Surg Oncol. 2019 Dec;26(13):4256-4263. doi: 10.1245/s10434-019-07725-w. Epub 2019 Aug 19. PMID 31429019